CLINICAL TRIAL: NCT03293355
Title: Multilevel Integration Strategies to Enhance Service Provider Networks in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Principal Investigator, Li Li, Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA041008 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2018-10

CONDITIONS: Linkage to Care
Keywords: People Living with HIV Who Use Drugs (PLHWUD); Community Health Workers (CHW); Multilevel Service Integration; HIV/AIDS; Vietnam
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care
- Intervention (Experimental): The VPN intervention has 2 in-person sessions:
  1) Providing training on service integration and team building for CHW and tools for them to network more effectively with OPC and MMT treatment providers as well as reach out to their patients; and 2) Learning to use effective communication tools such as motivational ruler and decision balance sheet to work more effectively with their patients and use Facebook group to facilitate collaboration among providers and e-chat for patient engagements. Sessions will occur once a week for two weeks, with each session featuring a different set of themes and relevant activities.
  Interventions: Behavioral: VPN

INTERVENTIONS:
Behavioral: VPN — Two in-person sessions will take place one week apart for the VPN intervention targeting CHW. The intervention contents aim to utilize traditional communications tools and the latest technology to tackle challenges faced by service providers working in commune health centers and the impact of these challenges on their patients' treatment initiation, retention, and adherence. In addition, booster sessions will be offered once every month during the first three months and once every three months thereafter. The booster sessions will focus on participants' reports of their experiences, reinforcement of efforts, and continued skill building for problem solving.
  Arms: Intervention

SUMMARY:
There is an urgent need for treatment service integration for People Living with HIV (PLH) because many PLH have comorbid conditions, including substance use disorders and psychiatric disorders, among others. Although providing integrated services to PLH who use drugs (PLHWUD) has been proven to produce positive outcomes, multilevel challenges must be addressed, including barriers at the policy, structural, and provider levels. Many countries, including Vietnam, face challenges in the pursuit of multilevel integration of combination treatment services and care. In Vietnam, injecting drug use accounts for nearly two-thirds of HIV infection, and methadone maintenance therapy (MMT) services have rapidly expanded to 135 clinics with over 25,000 clients since 2008. There is a timely call as well as an opportunity to identify, implement and evaluate new strategies to provide MMT and HIV treatment as an integrated service system for PLHWUD. The study will take advantage of this window of opportunity to explore and pilot integration strategies to address the multilevel challenges associated with service integration in Vietnam.

DETAILED DESCRIPTION:
The purpose of this study is to develop and pilot test intervention strategies at the provincial level (Aim 1), treatment agency level (Aim2), and community level (Aim 3). These strategies aim to strengthen both horizontal and vertical collaboration and networking among providers to better serve people living with HIV who use drugs (PLHWUD), including those who are already in treatment and those who need to be linked to service. Commune health workers (CHW) have great potentials to be mobilized to engage PLHWUD living in the community and to work with providers at treatment clinics to support PLHWUD treatment retention and adherence. E-technologies such as Facebook and e-chat will also be utilized to enhance provider-provider coordination and provider-patient interaction.

The Specific Aims of the study are as follows:

Aim 1: Develop and implement structural-level strategies by establishing a provincial coordination team to improve coordination and service integration.

Aim 2: Assess agency-level intervention outcomes on treatment-provider collaboration and service integration of OPC services and MMT programs.

Aim 3: Assess community provider-level intervention outcomes by evaluating whether: 1) CHW in the intervention group, compared to those in the control group, demonstrate improved levels of collaboration with other clinical agencies, communication with patients, and service referrals, and 2) PLHWUD in the intervention group, compared to those in the control group, demonstrate improvements in treatment initiation, retention and adherence, and other mental and biological outcomes.

Based on the findings from Aims 1 and 2 activities, this intervention will be conducted in four provinces of Vietnam(Bac Giang, Hai Duong, Nam Dinh, and Nghe An). Randomization will occur at the community level (20 communes assigned to the intervention group; 20 communes assigned to the control group).

CONTROL COMMUNE ACTIVITIES:

A total of 40 CHW from 20 communes assigned to the control group will be invited to participate in a one-time didactic lecture/meeting with other co-workers from their commune health centers to learn about the importance of service integration.

CHW(n=40) and PLHWUD(n=120) from the control commune health centers will participate in a baseline assessment and follow-up assessments at 3, 6, 9, 12-months.

INTERVENTION COMMUNE ACTIVITIES:

A total of 40 CHW from 20 communes assigned to the intervention group will be invited to participate in the intervention that will consist of two in-person sessions lasting approximately 90 minutes over two weeks with 8-10 CHW in each session.

Booster sessions of the intervention training will be offered to CHW once every month during the first three months and once every three months thereafter. The booster session will focus on CHW' reports of their experiences, reinforcement of efforts, and continued skill building for problem solving. CHW(n=40) and PLHWUD(n=120) from the intervention commune health centers will participate in a baseline assessment and follow-up assessments at 3, 6, 9, 12-months.

The efficacy of the intervention will be assessed at baseline, 3, 6, 9, and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

CHW:

* Age 18 or over
* Be a service provider to PLHWUD attending commune health centers in one of the 40 communes selected selected for the study
* Voluntary written informed consent

PLHWUD:

* Age 18 or over
* HIV positive (self-report)
* Currently using opiates or has a history of opiate use (self-report) and seeking services at the commune health centers in one of 40 communes selected from the study
* Has not received treatment services from OPC or MMT clinics (i.e., is treatment naive).
* Voluntary written informed consent

Exclusion Criteria:

CHW:

* Inability to give informed consent

PLHWUD:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
PLHWUD's service utilization | Changes from baseline to 3-, 6-, 9- and 12- month follow-ups
  This will be measured by PLHWUD's utilization of health services including OPC and MMT. Both their access and adherence to treatments will be assessed.
CHW interaction with providers of other treatment agencies | Changes from baseline to 3-, 6-, 9- and 12- month follow-ups
  This will be measured by a multi-item scale on interaction with other treatment providers

SECONDARY OUTCOMES:
PLHWUD's service satisfaction | Changes from baseline to 3-, 6-, 9- and 12- month follow-ups
  PLHWUD's service satisfaction will be measured using a 12-item scale to evaluate patients' service satisfaction with MMT and OPC treatment based on the Texas Christian University Client Evaluation of Self and Treatment (TCU-CEST) forms.
CHW's patient-provider interaction with PLHWUD | Changes from baseline to 3-, 6-, 9- and 12- month follow-ups
  CHW's communication and interaction with PLHWUD will be measured by a self-reported scale and the provider-patient communication logs.
CHW's service provision | Changes from baseline to 3-, 6-, 9- and 12- month follow-ups
  Service provision such as patient referrals will be captured by the reported frequency and type of service referrals made in the past three months to other treatment clinics will also be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, PhD, Principal Investigator — University of California, Los Angeles
Locations (4):
- Vietnam (4):
  - Commune Health Centers, Hải Dương, Hải Dương
  - Commune Health Centers, Nghi An, Nghệ An Province
  - Commune Health Centers, Bắc Giang
  - Commune Health Centers, Nam Định